CLINICAL TRIAL: NCT04044092
Title: Effects of Elongation Longitudinaux Avec Decoaption Osteo-Articulaire (ELDOA) in Cervical Disc Protrusion
Brief Title: Elongation Longitudinaux Avec Decoaption Osteo-Articulaire (ELDOA) in Cervical Disc Protrusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Muhammad Safdar Ch
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Cervical Disc Herniation
Keywords: Cervical Disc Protrusion; ELDOA,; Neck Pain; Neck Disability
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative physical therapy (Active Comparator): Moist hot packs, TENS, Cervical Traction, Neural Mobilization, Cervical Spine strengthening exercises
  Interventions: Other: Conservative physical therapy
- ELDOA stretching exercise (Experimental): ELDOA stretching exercise protocol along with Conservative physical therapy
  Interventions: Other: ELDOA stretching exercise

INTERVENTIONS:
Other: Conservative physical therapy — Moist hot packs, TENS, Cervical Traction, Neural Mobilization on alternate days Cervical Spine strengthening exercises 10 repetitions×1 set, 4 days/week. Total of 4 sessions were given each consisting of 40 mins.
  Arms: Conservative physical therapy
Other: ELDOA stretching exercise — Experimental group was given ELDOA stretching exercise protocol along with the moist hot packs, TENS, Cervical Traction, and Neural Mobilization on alternate days Cervical Spine strengthening exercises 10 repetitions×1 set, 4 days/week. Total of 4 sessions were given each consisting of 40 mins.
  Arms: ELDOA stretching exercise

SUMMARY:
The aim of this research is to find and compare the effect of conventional physical therapy and ELDOA stretching exercise on pain, range of motion and disability in patients with cervical disc protrusion. The Randomized controlled trials done at Armed Forces Institute of Rehabilitation Medicine, Rawalpindi. The sample size was 20. The subjects were divided in two groups, 10 subjects in conventional physical therapy group and 10 in ELDOA stretching exercise group. Study duration was of 6 months. Sampling technique applied was Convenient Sampling technique randomization in group through Lottery method (sealed envelope). Only 30-60 years individuals with cervical disc protrusion were included. Tools used in the study were measurement of ROM by bubble inclinometer, Numeric pain rating scale (NPRS) and neck disability index (NDI). Data was analyzed using SPSS 21.

DETAILED DESCRIPTION:
Cervical disc protrusion is a significant cause of neck and arm pain and disability in majority of individuals. It causes a great burden on physical, social and emotional quality of life of patients. The cervical disc protrusion is characterized by prolapsed nuclear material through the annulus into the spinal canal. The local mechanical or chemical irritation of neural structures typically leads to symptoms of radiculopathy, head and neck pain or myelopathy. The disc protrusion may be postero-central to compress the dura matter, causing multi segmental pain and affect the scapular area. It can also be postero-lateral causing the root signs, which have dermatomal behavior and affect the upper limb in specific pattern. Postero-central protrusion can also shift to postero-lateral with symptoms shifting from centralization to radiculopathy.

Symptomatic disc protrusions can occur at any age but have different clinical features depending on the age group. In young adults nucleus pulposus can involve which is rare in old age. Diagnoses can be established on clinical findings along with patient's history, the functional examination and MRI. Disc protrusion can occur in postero-central, lateral and Postero- lateral directions.

Movement of the disc posteriorly causes stress on the posterior longitudinal ligament and also on the anterior part of the Dura mater. As a result of this the pain travels in more than one segment with dural reference. This typical postero central protrusion causes the pain symptoms centrally and bilaterally. Postero lateral disc protrusion may irritate the nerve root, which causes a Segmental or root pain and paraesthesia. The goal of treatment in disc protrusion problems is to stop the conflict between the displaced disc material and affecting sensitive structure. Protruded disc fragment may affect the Dura matter, nerve roots and intervertebral joints.

ELDOA is a series of stretching exercises and body movements that uses the Centre of gravity and localizes a target area of the spine that need to be mobilized or re aligned by placing and maintaining tension on the fascia. In ELDOA improvement in the tone of the intrinsic muscles of the spine combined with reinforcing the extrinsic muscles related to the spine in the neck. The stretching of the interlinking Para spinal muscles and finally inter independent movement of "Junghans functional unit" is facilitated and it is emphasized that micro movement affects macro function. The basic working principle during an ELDOA stretching consists of creating a position that will target a specific segment i.e. the functional unit. The inferior segment is fixed while the superior segment is mobilized. The position is created in such to place all the inferior and superior myofascial chains under tension. The effects of ELDOA include decompression of the superior and inferior facet joints, allowing for more space, joint play, and the range of motion.

Except ELDOA the other different treatment methods for intervertebral disc protrusion includes the application of physical modalities, mechanical traction, specific physical therapeutic exercise, oral anti-inflammatory medication, and patient education. Disc decompression therapy, surgery, minimally invasive Oxygen- Ozone therapy that exploits the biochemical properties of a gas mixture of Oxygen and Ozone and administration of periganglionic injection of corticosteroid and an anesthetic agent.

Physiotherapy treatment protocol for cervical disc protrusion includes cervical traction, neural mobilization and cervical spine strengthening exercises to relieve stress on the muscles. ELDOA stretching exercise is a systematic technique that causes decompression of the superior and inferior facets of the involved segment, allowing for more space, joint play, and the range of motion. This study hypothesize that there is a difference between the effects of conventional physical therapy treatment and ELDOA stretching exercise for the disc protrusion. The objective of this study is to find the effects of ELDOA stretching technique and to compare it with conventional physical therapy treatment in patients with cervical disc protrusion.

Literature review A systematic and evidence based search of relevant literature was performed by utilizing PubMed and Google Scholar as search engines.

Search term for the initial literature review was disc protrusion, prevalence of neck pain, causes of neck pain, pathophysiology of disc protrusion, treatment options for disc protrusion, effects of ELDOA in disc protrusion. The search was limited to papers in English preferably published since 2000 with full text available. Different studies were available regarding cervical manipulation and its effects but limited data was available regarding the effects of ELDOA on cervical disc protrusion in recent years.

In 2016,The prevalence of playing related injuries in collegiate violinists and the physical, emotional, and mental effects of ELDOA. Conducted an exploratory study to investigate the effects of ELDOA on the perceived pain in collegiate violinists at Jacob School of Music Indiana University. The study findings were overall decrease in pain and some study participants indicated the physical, emotional, and mental benefits after doing ELDOA exercises such as improve body posture, increase flexibility, mobility, and range of motion. Participants also noticed a change in mental behavior as decrease in stress, anxiety, improved sleep patterns and some participants did not observed as much emotional or mental benefits as others.

Quasi experimental short time study on Fascia Stretching Improve the Pain and Functional Level in Disc Protrusion Patients: JRCRS; 2016. The study participants were administered ELDOA exercises with conservative physical therapy treatment in both cervical and lumbar disc protrusions. The result of this study showed that ELDOA has significant result to decrease pain and improved functional status of the subjects. The pre and post-treatment frequency and intensity of pain showed significant differences.

In a study on incidence of intervertebral disc protrusion disclosed by postmortem radiography and myelography, 60 % of patients over the age of 30 years have multiple anterior and lateral disc protrusion of witch 40% were posterior disc protrusions.

ELIGIBILITY:
Inclusion Criteria:

* MRI with grading of disc protrusion
* Radiculopathy
* Limited ROM (measured by bubble Inclinometer)
* Pain more than 3 on NPRS

Exclusion Criteria:

* Malignancy,
* Infection,
* Trauma,
* Bone deformities,
* Severe osteoporosis
* With marked bony and soft tissue disease
* Taking other treatment in the same period of the research

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Neck disability index | 4th day
  Changes from base line: Northwick disability index was developed first in Northwick Park hospital, England. It was designed to measure the neck pain and disability over time. It consists of 10, five parts sections. At the end, score is calculated by dividing the obtained score by total (50) multiplied by 100. As the driving section was missing in most of the female patients, total score was considered as 45 instead of 50.
Numeric Pain rating scale (NPRS) | 4th day
  Changes from base Line: Numeric Pain rating scale is a scale for pain starting from 0-10, where 0 indicate no pain and 10 indicate worst possible pain.
ROM Cervical Spine (Flexion) | 4th day
  Changes from the Baseline ROM: Range of Motion of Cervical spine flexion was taken with the help of bubble inclinometer
ROM Cervical Spine (Extension) | 4th day
  Changes from the Baseline ROM: Range of Motion of Cervical spine extension was taken with the help of bubble inclinometer
ROM Cervical Spine (Right side flexion) | 4th day
  Changes from the Baseline ROM: Range of Motion of Cervical spine right side flexion was taken with the help of bubble inclinometer
ROM Cervical Spine (Left side Flexion) | 4th day
  Changes from the Baseline ROM: Range of Motion of Cervical spine left side flexion was taken with the help of bubble inclinometer
ROM Cervical Spine (Right rotation) | 4th day
  Changes from the Baseline ROM: Range of Motion of Cervical spine right rotation was taken with the help of bubble inclinometer
ROM Cervical Spine (Left rotation) | 4th day
  Changes from the Baseline ROM: Range of Motion of Cervical spine left rotation was taken with the help of bubble inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Risbud MV, Shapiro IM. Role of cytokines in intervertebral disc degeneration: pain and disc content. Nat Rev Rheumatol. 2014 Jan;10(1):44-56. doi: 10.1038/nrrheum.2013.160. Epub 2013 Oct 29. PMID 24166242
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Schoenfeld AJ, George AA, Bader JO, Caram PM Jr. Incidence and epidemiology of cervical radiculopathy in the United States military: 2000 to 2009. J Spinal Disord Tech. 2012 Feb;25(1):17-22. doi: 10.1097/BSD.0b013e31820d77ea. PMID 21430568
- [Background] Gross AR, Hoving JL, Haines TA, Goldsmith CH, Kay T, Aker P, Bronfort G; Cervical Overview Group. A Cochrane review of manipulation and mobilization for mechanical neck disorders. Spine (Phila Pa 1976). 2004 Jul 15;29(14):1541-8. doi: 10.1097/01.brs.0000131218.35875.ed. PMID 15247576
- [Background] Bronfort G, Haas M, Evans RL, Bouter LM. Efficacy of spinal manipulation and mobilization for low back pain and neck pain: a systematic review and best evidence synthesis. Spine J. 2004 May-Jun;4(3):335-56. doi: 10.1016/j.spinee.2003.06.002. PMID 15125860
- [Background] Hammer WI. Functional soft-tissue examination and treatment by manual methods: Jones & Bartlett Learning; 2007. 689-690
- [Background] Sajjad AG KA. Fascia Stretching Improve the Pain and Functional Level in Disc Protrusion Patients: Journal of Riphah College of Rehabilitation Sciences; 2016.